CLINICAL TRIAL: NCT03173131
Title: Opioid Consumption After Orthopaedic Surgery: Prospective Randomized Trial on the Effects of Pre-Operative Counseling
Brief Title: Opioid Consumption After Orthopaedic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 17D.131
Record Dates: First submitted 2017-05-05; First posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid counseling group (Experimental): Counseling provided to patients prior to surgery regarding opioid usage, side effect, long term effect and risks of opioids.
  Interventions: Behavioral: Pre-operative opioid counseling
- No Counseling (No Intervention): No preoperative counseling will be provided to this group. Standard medication information will be provided only.

INTERVENTIONS:
Behavioral: Pre-operative opioid counseling — Patients will be randomized to receive counseling regarding opioid medication and post operative pain control.
  Arms: Opioid counseling group

SUMMARY:
This is a randomized controlled study that will involve fellowship-trained board certified orthopaedic surgeons in four different subspecialties (hand surgery, sports surgery, shoulder and elbow surgery, and foot and ankle surgery) within our practice group. Consenting patients will be randomized to the treatment group (receiving preoperative counseling) or to the control group (no preoperative counseling). The control limb will provide us with information regarding average opioid consumption following common outpatient orthopedic procedures, and the study limb will allow us to evaluate the effect of the pre-operative opioid counseling.

DETAILED DESCRIPTION:
Over the past two decades in the United States, the opioid epidemic has escalated at a startling rate and prescription opioids are a large contributor to this problem. Studies show that there is an excessive amount of opioids being prescribed for orthopedic procedures. An accurate understanding of opioid consumption following common outpatient orthopedic surgery is imperative in order to treat pain appropriately relative to the surgery being performed without leading to excess narcotic prescribing.

The purpose of the study is threefold: to better understand typical opioid consumption following common outpatient orthopedic surgeries, to generate prescribing guidelines to optimize opioid prescribing, and to understand the effect of pre-operative opioid counseling on opioid consumption following these procedures.

This is a prospective randomized controlled study that will involve eight fellowship-trained board certified orthopaedic surgeons in four different subspecialties (hand surgery, sports surgery, shoulder and elbow surgery, and foot and ankle surgery). Consenting patients will be randomized to the treatment group (receiving preoperative counseling) or to the control group (no preoperative counseling). The control limb will provide us with information regarding average opioid consumption following common outpatient orthopedic procedures, and the study limb will allow us to evaluate the effect of the pre-operative counseling.

Basic demographic and surgical data will be collected. Primary outcomes will be assessed at the post-operative visit. These include the total number of opioid pills consumed, average daily pain scores, and adverse effects. Secondary outcomes include the number of days the medication was used, medication refill requests, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients indicated to undergo outpatient orthopedic surgery in one of the four areas included in the study (hand surgery, sports surgery, shoulder and elbow surgery, and foot and ankle surgery).
* Age eligibility is > 18 years of age.

Exclusion Criteria:

* Inpatient procedures.
* Pediatric patients (age < 18 years).
* Known allergy to narcotic medication.
* Pregnant female patients.
* Non-English speaking patients
* History of chronic pain and/or narcotic use preoperatively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2017-09-01 (Estimated); Study Completion 2017-10-01 (Estimated)

PRIMARY OUTCOMES:
Post operative opioid consumption | 3 months
  The primary outcome measure will be post operative opioid consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Asif Ilyas, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No